CLINICAL TRIAL: NCT03256578
Title: A Multi-center Randomized Controlled Trial of Respiratory Function Monitoring During Stabilization of Preterm Infants at Birth
Brief Title: Monitoring Neonatal Resuscitation Trial
Acronym: MONITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Leiden University Medical Center (Other); Royal Women's Hospital in Melbourne, Australia (Unknown); Maternal & Children's University Hospital, Valencia, Spain (Other); Vittore Buzzi Children's Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Foglia, Assistant Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 826695; NTR4104 (Registry Identifier: Netherlands Trial Registry)
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Resuscitation; Neonatal Prematurity; Positive-Pressure Respiration
Keywords: Resuscitation; Neonatal Prematurity; Positive-Pressure Ventilation; Respiratory Function Monitor

STUDY DESIGN:
Intervention Model Description: Eligible infants are either randomized to the intervention, where the clinical team will be able to directly observe the monitor or randomized to the RFM-masked display arm, where they will only see a black screen.
Who Masked: Outcomes Assessor
Masking Description: The waveform data and videos captured during the study intervention will be centralized to Leiden University Medical Center. The team at Leiden University Medical Center assessing the outcomes will be will be blinded to the randomization allocation of the infant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- RFM visible (Experimental): During resuscitation immediately following delivery the providers involved in the care of enrolled eligible infants can see the information displayed on the New Life Box Respiratory Function Monitor screen.
  Interventions: Device: New Life Box Respiratory Function Monitor
- RFM masked (No Intervention): During resuscitation immediately following delivery the providers involved in the care of enrolled eligible infants cannot see the information displayed on the New Life Box Respiratory Function Monitor screen. Though the display is masked, data is collected in the background.

INTERVENTIONS:
Device: New Life Box Respiratory Function Monitor — The intervention is the use of a visible New Life Box Respiratory Function Monitor display in infants born between 24 and 27 6/7 weeks gestation receiving PPV for resuscitation after birth.
  Arms: RFM visible

SUMMARY:
This is a randomized trial to determine if a visible respiratory function monitor (RFM) displaying realtime measurements of delivered inflations improves clinical providers ability to perform positive pressure ventilation (PPV) within a pre-defined target tidal volume in preterm infants after birth.

DETAILED DESCRIPTION:
Recently, it has been demonstrated that the use of a respiratory function monitor (RFM) can guide PPV in the DR.(Wood, Schmolzer) In this study, the New Life Box, (Advanced Life Diagnostics, Weener, Germany) a neonatal Respiratory Monitor (RFM), will be used to measure and calculate inflation pressures, flow, and tidal volumes in all enrolled infants. The New Life Box uses a small variable orifice anemometer to measure gas flow in and out of a face-mask or endotracheal tube. This signal is automatically integrated to provide inspired (Vti) and expired (Vte) tidal volume. The difference equals the leak from the facemask or endotracheal tube. Complete airway obstruction occurs when no flow of gas into or away from the infant is seen during a positive pressure inflation. The RFM can also calculate and measure respiratory rate and minute volume, inflations and spontaneous inspirations, and all ventilation pressures. Using customized software heart rate, oxygen saturation and expired carbon dioxide can be integrated into the RFM.

The NewLife Box monitor presents graphical information for pressure, flow, and volume. In addition, the monitor displays numeric data for pressure (PIP and PEEP), tidal volume (Vti, Vte), flow, respiratory rate and percent leak. The monitor integrates and displays physiologic data streaming from the patient (heart rate and oxygen saturation) as well as FiO2 from an oxygen analyzer in the inspiratory limb of the respiratory circuit. If enabled, the monitor can incorporate video captured from an external camera. The video serves as a helpful aid in the interpretation of the events during the RFM waveform recordings.

The use of an RFM in the DR has the potential to improve neonatal respiratory support and reduce lung injury.

The primary objective of this study is to test the hypothesis that observing the data and waveforms displayed on an RFM during the provision of PPV to preterm infants (24-27 6/7 weeks gestation) after birth will increase the proportion of inflations performed with a predefined VTe "safe range" of 4 - 8 mls/kg.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA) 24 - 27 6/7 weeks at birth, by best obstetrical
* Receive positive pressure ventilation during delivery room resuscitation

Exclusion Criteria:

* Known major anomalies including that may affect measured cardiorespiratory parameters: congenital diaphragmatic hernia, trachea-oesophageal fistula, cyanotic heart disease, pulmonary hypoplasia
* RFM not available during resuscitation

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjan te Pas, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood FE, Morley CJ, Dawson JA, Davis PG. A respiratory function monitor improves mask ventilation. Arch Dis Child Fetal Neonatal Ed. 2008 Sep;93(5):F380-1. doi: 10.1136/adc.2007.120097. Epub 2008 Jan 11. PMID 18192329
- [Background] Schmolzer GM, Kamlin OC, Dawson JA, te Pas AB, Morley CJ, Davis PG. Respiratory monitoring of neonatal resuscitation. Arch Dis Child Fetal Neonatal Ed. 2010 Jul;95(4):F295-303. doi: 10.1136/adc.2009.165878. Epub 2009 Sep 22. PMID 19776023
- [Derived] van Zanten HA, Kuypers KLAM, van Zwet EW, van Vonderen JJ, Kamlin COF, Springer L, Lista G, Cavigioli F, Vento M, Nunez-Ramiro A, Oberthuer A, Kribs A, Kuester H, Horn S, Weinberg DD, Foglia EE, Morley CJ, Davis PG, Te Pas AB. A multi-centre randomised controlled trial of respiratory function monitoring during stabilisation of very preterm infants at birth. Resuscitation. 2021 Oct;167:317-325. doi: 10.1016/j.resuscitation.2021.07.012. Epub 2021 Jul 22. PMID 34302924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between Oct 2013-May 2019 in 7 NICUs in 6 Countries (Netherlands, Australia, Germany, Spain, Italy, and the United States). IRBs at each site approved the study. At five of the seven non-US sites, deferred consent was endorsed for use when there was insufficient time for antenatal consent, or it was considered inappropriate.
Pre-assignment Details: Infants with antenatal enrollment into the trial were excluded from randomization if their delivery occurred outside of the gestational age eligibility window.Post-randomization exclusion occurred if postnatal consent was not obtained, no IPPV delivered, equipment failure, or a congenital anomaly was discovered.
Period: Overall Study
Arm/Group | RFM Visible | RFM Masked
Started | 204 | 206
Completed | 138 | 150
Not Completed | 66 | 56
Not completed — Excluded Post Randomization | 66 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RFM Visible | RFM Masked | Total
Number analyzed (Participants) | 138 | 150 | 288
Age, Customized [Median (Inter-Quartile Range); unit: weeks]
  Gestational age in weeks | 26 [25 to 27] | 26 [25 to 27] | 26 [25 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 67 | 131
  Male | 74 | 83 | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21
  Netherlands | 42 | 54 | 96
  Italy | 31 | 27 | 58
  Australia | 36 | 38 | 74
  Spain | 13 | 14 | 27
  Germany | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Positive-Pressure Ventilation Inflations Between 4 - 8 Mls/kg
Description: To test the hypothesis that observing the data and waveforms displayed on an RFM during the provision of PPV to preterm infants (24-27 6/7 weeks gestation) after birth will increase the percentage of inflations performed with a predefined VTe "safe range" of 4 - 8 mls/kg.
Time Frame: the first 15 minutes of resuscitation
Measure: Median (Inter-Quartile Range); unit: percentage of inflations
Units Other Than Participants: Total inflations
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Number analyzed (Total inflations) | 25432 | 25920
percentage of inflations | 30.2 [18.0 to 41.6] | 30.7 [15.8 to 43.4]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.896, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage of Oxygen Saturation (SpO2) in the First 5 Minutes of Life
Description: Median percentage of oxygen saturation (SpO2) captured on the Respiratory Function Monitor in the first 5 minutes of life
Time Frame: approximately first 5 minutes of life
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of oxygen saturation | 59 [46 to 71] | 63 [52 to 72]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.107, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Heart Rate in the First 10 Minutes of Life
Description: Median Heart rate captured on the Respiratory Function Monitor between 3 and10 minutes of life
Time Frame: between 3 and 10 minutes of life
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
beats per minute | 144 [130 to 156] | 143 [127 to 158]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.847, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Time With Mask Leak During PPV Ventilation
Description: Percentage of time with significant mask leak (defined as > 60%) during the duration of PPV ventilation per infant in the first 15 minutes of resuscitation.
Time Frame: approximately first 15 minutes of resuscitation
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of time | 17.4 [7.2 to 33.3] | 13.6 [3.7 to 32.1]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.126, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of PPV Inflations With Airway Obstruction
Description: Percentage of PPV inflations with airway obstruction in the first 15 minutes of resuscitation. Airway obstruction is defined as Vte <1 mL/kg, with minimal mask leak (<25%) during an inflation and flattening of the flow waves.
Time Frame: approximately first 15 minutes of resuscitation
Measure: Median (Inter-Quartile Range); unit: percentage of inflations
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of inflations | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.346, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage of PPV Inflations With Inadequate Tidal Volume
Description: Percentage of PPV inflations with inadequate tidal volume defined as Vte <4 ml/kg in the first 15 minutes of resuscitation.
Time Frame: approximately first 15 minutes of resuscitation
Measure: Median (Inter-Quartile Range); unit: percentage of inflations
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of inflations | 40.7 [20.5 to 62.4] | 34.1 [18.5 to 52.6]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.094, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Oxygen Saturation (SpO2) in the First 10 Minutes of Life
Description: Median percentage of Oxygen saturation (SpO2) captured on the Respiratory Function Monitor between 3 and 10 minutes of life
Time Frame: Between 3 and 10 minutes of life
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of oxygen saturation | 84 [74 to 89] | 85 [75 to 90]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.656, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Fraction of Inspired Oxygen (FiO2) Provided in the First 10 Minutes of Life
Description: Median fraction of inspired oxygen (FiO2) provided to the infant between 3 and 10 minutes of life
Time Frame: between 3 and 10 minutes of life
Measure: Median (Inter-Quartile Range); unit: percentage fraction of inspired oxygen
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage fraction of inspired oxygen | 51 [36 to 74] | 49 [36 to 69]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.434, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Total Duration With FiO2 of 100% Delivered in the First 10 Minutes of Life
Description: Total duration of time where FiO2 of 100% is delivered to the patient in first 10 minutes of life will be calculated taking into consideration birth weight, tidal volume, respiratory rate, FiO2 and timing of stabilization.
Time Frame: approximately first 10 minutes of life
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
percentage of time | 0 [0 to 13.2] | 0 [0 to 11.9]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.903, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Number of Participants Receiving Endotracheal Intubation in the Delivery Room
Description: Number of Participants receiving Endotracheal Intubation in the delivery room from time of birth to admission to NICU
Time Frame: from time of birth to admission to NICU
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Participants | 47 | 54
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.699, Chi-squared

11. Secondary Outcome: Number of Participants Requiring Inotropes for Circulatory Support
Description: Number of participants requiring inotropes for circulatory support in the Neonatal Intensive Care Unit in the first 3 days after birth
Time Frame: within the first 3 days after birth
Population: 1 infant in the RFM masked arm died in the delivery room and therefore did not have NICU data available to contribute to this secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 22 | 32
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.231, Chi-squared

12. Secondary Outcome: Number of Participants With Pneumothorax
Description: Number of participants with pneumothorax in the first 72 hours after birth reported by a radiologist masked to the intervention
Time Frame: in the first 72 hours after birth
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 6 | 11
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.283, Chi-squared; Risk Ratio (RR) = 0.593, 95% CI 2-sided [0.225 to 1.561]

13. Secondary Outcome: Number of Participants With Pulmonary Interstitial Emphysema
Description: Number of participants with Pulmonary Interstitial Emphysema in the first 72 hours after birth reported by a radiologist masked to the intervention
Time Frame: in the first 72 hours of life
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 12 | 7
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.168, Chi-squared; Risk Ratio (RR) = 1.864, 95% CI 2-sided [0.756 to 4.599]

14. Secondary Outcome: Number of Participants With Abnormal Cranial Ultrasound Findings
Description: Number of participants with abnormal cranial ultrasound findings (i) all intraventricular hemorrhage, (ii) severe - ie. Papile grade III and IV intraventricular hemorrhage, (iii) cystic periventricular leukomalacia through study completion, an average of 4 months
Time Frame: through study completion, an average of 4 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 36 | 58
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.024, Chi-squared; Risk Ratio (RR) = 0.670, 95% CI 2-sided [0.474 to 0.947]

15. Secondary Outcome: Duration of Endotracheal Ventilation
Description: Duration of endotracheal (ET) ventilation days through study completion, an average of 4 months
Time Frame: days through study completion, an average of 4 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
days | 7 [1 to 20] | 6 [1 to 17]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.585, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Duration of Non-invasive Ventilation
Description: Duration of non-invasive ventilation, days through study completion, an average of 4 months
Time Frame: days through study completion, an average of 4 months
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
days | 41 [29 to 56] | 37 [16 to 55]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.342, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Duration of Supplemental Oxygen Therapy
Description: Duration of supplemental oxygen therapy days through study completion, an average of 4 months
Time Frame: days through study completion, an average of 4 months
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
days | 43 [15 to 77] | 35 [8 to 75]
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.431, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Total Duration of Assisted Ventilation
Description: Total duration of assisted ventilation (ET, CPAP) in hours through study completion, an average of 4 months
Time Frame: through study completion, an average of 4 months
Population: Outcome measure was not analyzed as the way the data was collected did not allow for a total calculation of all assisted ventilation. (Data collected at all centers provided the data in days (defined as minimum of 6 hours per day) separately for mechanical and non-invasive ventilation, therefore even a total estimation in days may not be representative).
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With a Diagnosis of Bronchopulmonary Dysplasia
Description: Number of participants with a diagnosis of bronchopulmonary dysplasia (BPD) at 36 weeks corrected gestational age defined as the need for supplementary oxygen and/or any form respiratory support
Time Frame: at 36 weeks corrected gestational age
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants
  Mild | 32 | 26
  Moderate | 8 | 10
  Severe | 30 | 41
  No BPD | 68 | 72
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.518, Chi-squared; Risk Ratio (RR) = 1.059, 95% CI 2-sided [0.854 to 1.313]

20. Secondary Outcome: Neonatal Mortality
Description: Neonatal mortality from the time of birth until hospital discharge or 44 weeks corrected gestational age, whichever occurred first
Time Frame: from time of birth until discharge from hospital, up to 44 weeks corrected gestational age
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Participants | 21 | 24
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.855, Chi-squared; Risk Ratio (RR) = 0.951, 95% CI 2-sided [0.555 to 1.629]

21. Secondary Outcome: Composite Outcome of Death or BPD
Description: Composite outcome of death or BPD. BPD assessed at corrected gestational age of 36 weeks; death assessed from time of birth until discharge, up to 44 weeks corrected gestational age
Time Frame: BPD assessed at corrected gestational age of 36 weeks; death assessed from the time of birth until hospital discharge or 44 weeks corrected gestational age, whichever occurred first
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Participants | 84 | 96
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.524, Chi-squared; Risk Ratio (RR) = 0.994, 95% CI 2-sided [0.834 to 1.186]

22. Secondary Outcome: Number of Participants With Retinopathy of Prematurity Requiring Treatment
Description: Number of participants with Retinopathy of prematurity requiring treatment before hospital discharge, an average of 4 months
Time Frame: before hospital discharge, an average of 4 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 9 | 15
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.280, Chi-squared; Risk Ratio (RR) = 0.649, 95% CI 2-sided [0.294 to 1.434]

23. Secondary Outcome: Number of Participants With a Diagnosis of Necrotizing Enterocolitis
Description: Number of participants with a diagnosis of Necrotizing enterocolitis grade 2 or more before hospital discharge, an average of 4 months
Time Frame: before hospital discharge, an average of 4 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 17 | 13
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.339, Chi-squared; Risk Ratio (RR) = 1.393, 95% CI 2-sided [0.703 to 2.760]

24. Secondary Outcome: Number of Participants Requiring Fluid Boluses for Circulatory Support
Description: Number of participants requiring fluid boluses for circulatory support in the Neonatal Intensive Care Unit within the first 3 days of life
Time Frame: within the first 3 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 149
Participants | 36 | 45
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.486, Chi-squared

25. Secondary Outcome: Number of Participants With Endotracheal Intubation in the NICU
Description: Number of Participants with Endotracheal Intubation in the NICU in the first 24 hours of life
Time Frame: in the first 24 hours of life
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Participants | 26 | 30
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 0.655, Chi-squared

26. Secondary Outcome: Neonatal Mortality in the Delivery Room
Description: Neonatal Mortality in the delivery room from time of birth until transfer to NICU
Time Frame: from time of birth until transfer to NICU
Measure: Count of Participants; unit: Participants
Arm/Group | RFM Visible | RFM Masked
Number analyzed (Participants) | 138 | 150
Participants | 0 | 1
Statistical Analysis 1: Comparison: RFM Visible vs RFM Masked; Test type: Superiority; p = 1.00, Chi-squared; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.99 to 1.02]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of birth (in the delivery room) to the time of transfer to the Neonatal Intensive Care Unit. All cause mortality was documented from the time of birth until hospital discharge or 44 weeks corrected gestational age, whichever occurred first.
Description: Need for positive pressure after birth is an inclusion criterion for this study, therefore respiratory failure requiring PPV or endotracheal intubation after birth was not considered an adverse event.
Arm/Group | RFM Visible | RFM Masked
All-Cause Mortality (participants affected / at risk) | 21/138 | 24/150
Serious Adverse Events (participants affected / at risk) | 3/138 | 4/150
Other Adverse Events (participants affected / at risk) | 0/138 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RFM Visible (N=138) | RFM Masked (N=150)
Chest Compressions (Respiratory, thoracic and mediastinal disorders) | 2 | 3 — Chest Compressions during neonatal resuscitation in the delivery room
Adrenaline (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Adrenaline during neonatal resuscitation in the delivery room

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03256578/Prot_SAP_002.pdf
  • Informed Consent Form (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03256578/ICF_003.pdf